CLINICAL TRIAL: NCT05855746
Title: Colchicine Versus Placebo in Acute Myocarditis Patients to Reduce Late Gadolinium Enhancement Mass on Cardiac Magnetic Resonance and the Risk of Clinical Outcomes: The ARGO Trial
Brief Title: Colchicine Versus Placebo in Acute Myocarditis Patients
Acronym: ARGO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hospices Civils de Lyon (Other); Fonds de Dotation ACTION (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP211429
Record Dates: First submitted 2023-04-21; First posted 2023-05-11 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocarditis
Keywords: Myocarditis; Inflammation; Colchicine
MeSH Terms: conditions — Myocarditis; Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: This is a prospective, two arms, randomized (1:1), double blind, superiority study evaluating colchicine versus placebo administrated during six months among participants with acute myocarditis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Participant receive in addition to standard of care therapy, six months of Colchicine
  Interventions: Drug: Colchicine Pill
- Placebo (Placebo Comparator): Participant receive in addition to standard of care therapy, six months of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine Pill — Participant receive, in addition to standard of care therapy, six months of colchicine (at a dose of 0.5 mg twice daily, morning and evening) beginning maximum 72 hours post-randomization. The standard of care is defined according to the European consensus paper as follow: All participants without contraindication receive a betablockers, and heart failure ESC (European Society of Cardiology) guidelines directed medical therapies if LVEF < 50% (Left Ventricular Ejection Fraction), including ACE (Angiotensin-Converting Enzyme) inhibitors, diuretics if indicated. The choice of the dosage and the drug is left at the investigator decision.
  During the six months of the treatment administration, in case of severe adverse reaction (such as nausea and/or diarrhea during five days), a dose reduction could be considered by the investigator: half of the study protocol dose could be accepted (0.5 mg per day in the morning). In case of remaining adverse reactions, the study drug should be stopped.
  Other Names: Colchicine
  Arms: Colchicine
Drug: Placebo — Participant receive, in addition to standard of care therapy, six months of placebo (at a dose of 0.5 mg twice daily, morning and evening) beginning maximum 72 hours post-randomization.
  The standard of care is defined according to the European consensus paper as follow: All participants without contraindication receive a betablockers, and heart failure ESC (European Society of Cardiology) guidelines directed medical therapies if LVEF < 50% (Left Ventricular Ejection Fraction), including ACE (Angiotensin-Converting Enzyme) inhibitors, diuretics if indicated. The choice of the dosage and the drug is left at the investigator decision.
  Arms: Placebo

SUMMARY:
Myocarditis is an inflammatory disease of the heart, mostly caused by viruses. Patients with acute myocarditis are exposed to several complications: recurrence, ventricular arrhythmias (from 5 to 30%), heart failure (5-10%), death or heart transplantation (< 4%). To date, there is no specific treatment for myocarditis. Patient management only focuses upon empirical optimal care of arrhythmia and heart failure.

There is a strong rationale for using colchicine in acute myocarditis:

* the IL1 (Interleukin1) pathway plays a detrimental role in acute myocarditis. NLRP3 (NOD-like receptor family, pyrin domain containing 3) inflammasome assembly, and subsequent IL-1beta production, are profoundly inhibited by colchicine.
* colchicine has been shown to improve cardiac outcomes in inflammatory cardiac disorders, including pericarditis, coronary artery disease, and post pericardiotomy syndrome.
* In murine model of CVB3-induced myocarditis (coxsackievirus B3), colchicine improved myocarditis through reduction of NLRP3 activity.
* Small case series with improvement of left ejection fraction in myocarditis following low-dose colchicine in addition to conventional heart failure therapy have been reported.

With its pleiotropic anti-inflammatory effect in the pro-inflammatory cascade, reducing the myocardial damage and cell death induced during myocarditis, colchicine has the potential to reduce the risk of heart failure and ventricular arrhythmias. Finally, colchicine is a drug widely available, at low cost, and has a long and well-known safety record.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multicenter, double blind, controlled versus placebo, phase III study in which two groups of participants are compared: a group treated with the experimental treatment Colchicine (in addition to standard of care therapy) compared to a control group that receive the corresponding placebo (in addition to standard of care therapy).

The inclusion visit takes place during the initial hospitalization stay. The study is presented to all patients presenting with acute myocarditis symptoms and inclusion criteria, hospitalized in participating centers.

Once eligible participants have been informed and signed their informed consent, they are randomized (1:1) by a centralized web system (IWRS) in the experimental group (Colchicine) or the control group (Placebo).

Participants receive then a numbered box with three months' treatment of Colchicine or placebo. The treatment must start at least within 72h after randomization. Another dispensing is performed during the three months' follow-up visit.

All randomized participants are followed during six months after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptom onset of 21 days or less,
* Chest pain and/or Heart failure symptoms and/or palpitations
* Troponins superior to 99 percentile of reference value,
* Myocarditis diagnostic confirmation (by Contrast-Enhanced Cardiac Magnetic Resonance (CMR), according to the Lake Louise criteria (2009 or later),
* No evidence for ischemic heart disease on coronary angiography or coronary computed tomography angiography for patients with age superior to 40-year-old with one or more cardiovascular risk factor (hypertension, smoking, hypercholesterolemia, diabetes, personal or family history of coronary artery disease),
* Woman of child-bearing age with an effective contraception method according to the investigator for the duration of treatment and one month after,
* Man accepting effective contraception for the duration of treatment and one month after,
* Participant with affiliation to the French Health Care System "sécurité sociale",
* Written informed consent of the patient obtained.

Exclusion Criteria:

* Cardiogenic shock requiring inotropes or vasopressors (patients with inotropes discontinued for more than 24 hours can be enrolled)
* Giant cell myocarditis or eosinophilic myocarditis
* Acute coronary syndrome or known coronary stenosis superior to 50%
* Toxic cardiomyopathy
* Active chronic inflammatory disease, chronic active infection, evolving cancer
* A recent severe sepsis (7 days)
* Hypersensitivity to Investgational Medical Product's active substances (colchicine) or to any of the excipients (including lactose, sucrose, microcrystalline cellulose, colloidal silica, magnesium stearate, colourants : E127, Dual Red 40 )
* Any known contra-indication to CMR or associated contract products (claustrophobia; intra-ocular metal foreign bodies, clips such as cerebral, carotid, or aortic aneurysm, cochlear implants, any implant held in by magnet, non-MR compatible cardiac devices (pace maker or defibrillator); history of hypersensitivity to gadoteric acid or to gadolinium contrast agents or to meglumine),
* Chronic treatment with corticosteroids or Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) or immunosuppressant.
* Sarcoidosis
* Severe liver (Child Pugh C) or known renal dysfunction (known Glomerular Filtration Rate (GFR) less or equal to 30 ml/min according Cockroft),
* Cytopenia : hemoglobin less than 100 grams/L, white blood cell count less than 3.0 G/L, platelet count less than 100 G/L
* Major digestive disorders (chronic diarrhea, inflammatory disease of the digestive tract as uncontrolled ulcerative colitis or active Crohn disease)
* Immunosuppression, spinal cord aplasia
* Hemopathy
* Hypereosinophilia more than 0.5 G/L
* Pregnant or nursing women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive local laboratory test,
* Administration of any investigational drug or participation in another interventional trial, within 30 days before randomization,
* Participant under treatment having an interaction with colchicine [macrolides (telithromycin, azithromycin, clarithromycin, dirithromycin, erythromycin, josamycin, midecamycin, roxithromycin), pristinamycin,, cyclosporine, verapamil, all protease inhibitors, telaprevir, CYP3A4 powerful inhibitors, azole antifungals, vitamin K antagonists]
* Participant under legal protection: under guardianship (trusteeship or curatorship)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-01-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Extent of Late Gadolinium Enhancement (LGE) evaluated on Cardiac Magnetic Resonance (CMR) | Six months post-randomization
  Extent of LGE (pourcentage of left ventricle mass) is evaluated (centralized reading by the Corelab) on CMR performed at six months and compared to baseline CMR (performed at the hospital admision or inclusion).
  The inclusion visit takes place during the initial hospitalization.
Composite Clinical primary outcome | Six months post-randomization
  Composite Clinical primary outcome is assessed during the study period at six months on:
  * the rate of heart Failure or acute myocarditis recurrence;
  * or the rate of clinically relevant chest pain (defined as leading to an unplanned/urgent consultation or hospitalization or requiring an additional treatment);
  * or the rate of sustained ventricular arrhythmias;
  * or the rate of left ventricular assistance;
  * or the rate of heart transplantation;
  * or the rate of cardiovascular death

SECONDARY OUTCOMES:
Safety of colchicine | Six months post-randomization
  Safety of colchicine is defined as :
  * Rate of Serious Adverse Events related to colchicine
  * Rate of permanent treatment discontinuation
  * Rate of diarrhea
  * Rate of nausea and/or vomiting
  * Rate of myelotoxicity (evaluated on Complete Blood Count)
  * Renal function evaluated by creatinine level and creatinine clearance (MDRD)
Composite clinical secondary outcome | one year post-randomization
  Composite Clinical secondary outcome is assessed during the study period at one year on:
  * Rate of heart failure or acute myocarditis recurrence
  * Rate of clinically relevant chest pain (defined as leading to an unplanned/urgent consultation or hospitalization or requiring an additional treatment)
  * Rate of sustained ventricular arrhythmias
  * Rate of left ventricular assistance or heart transplantation
  * Rate of cardiovascular death
Rate of heart failure at 6 months | Six months post-randomization
  Rate of heart failure is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of acute myocarditis recurrence at 6 months | Six months post-randomization
  Rate of acute myocarditis recurrence is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of clinically relevant chest pain at 6 months | Six months post-randomization
  Rate of clinically relevant chest pain (defined as leading to an unplanned/urgent consultation or hospitalization or requiring an additional treatment) is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of sustained ventricular arrhythmias at 6 months | Six months post-randomization
  Rate of sustained ventricular arrhythmias is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of left ventricular assistance at 6 months | Six months post-randomization
  Rate of left ventricular assistance is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of heart transplantation at 6 months | Six months post-randomization
  Rate of heart transplantation is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of cardiovascular death at 6 months | Six months post-randomization
  Rate of cardiovascular death is a component of the composite clinical secondary endpoint. It is assessed at 6 months.
Rate of heart failure at 1 year | One year post-randomization
  Rate of heart failure is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Rate of acute myocarditis recurrence at 1 year | One year post-randomization
  Rate ofacute myocarditis recurrence is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Rate of clinically relevant chest pain at 1 year | One year post-randomization
  Rate of clinically relevant chest pain (defined as leading to an unplanned/urgent consultation or hospitalization or requiring an additional treatment) is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Rate of sustained ventricular arrhythmias at 1 year | One year post-randomization
  Rate of sustained ventricular arrhythmias is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Rate of left ventricular assistance at 1 year | One year post-randomization
  Rate of left ventricular assistance is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Rate of heart transplantation at 1 year | One year post-randomization
  Rate of heart transplantation is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Rate of cardiovascular death at 1 year | One year post-randomization
  Rate of cardiovascular death is a component of the composite clinical secondary endpoint. It is assessed at 1 year.
Left ventricular volume on Cardiac Magnetic Resonance (CMR) | Six months post-randomization
  Left Ventricular Ejection Fraction (LVEF), left ventricular end-diastolic and left ventricular end-systolic volumes are evaluated (centralized reading by the Corelab) on CMR performed at six months and compared to baseline CMR (performed at the hospital admision or inclusion).
Left ventricular volume on transthoracic echocardiography (TTE) | 6 months post-randomization
  Relative variation in Left ventricular ejection fraction (LVEF), end-diastolic volume and end-systolic volume between baseline and 6-months as determined by TTE.
Relative variation in Extent of late gadolinium enhancement (LGE) and edema | Six months post-randomization
  Relative variation in LGE and edema between baseline and six months determined centrally by the Corelab on the CMR
Tissue properties evaluated on Cardiac Magnetic Resonance (CMR) | Six months post-randomization
  Cardiac magnetic resonance criteria: value of native T1 and T2 mapping (ms), pourcentage of extracellular volume
Serum biomarkers | Six months post-randomization
  Serum biomarkers at hospital admission, 24h and 48h (after admission) and at six months: Troponin (I or T according to investigator), N-terminal pro-brain natriuretic peptide (NT-pro BNP), C-Reactiv Protein (CRP) and Creatin Kinase (CK)
Specific Inflammatory markers | Six months post-randomization
  Analysis of specific Inflammatory markers only for participating centers of biocollection at six months post-randomization versus baseline (inclusion; 24 hours and 48 hours post-inclusion) : interleukin 6 (IL-6), interleukin 1 beta (IL-1bβ) and ST2 (or soluble interleukin 1 receptor-like 1). Patients undergo two blood samples of 4 mL at inclusion ; 24 hours and 48 hours after the inclusion visit, if the patient is still in hospital; and at 6 months post-randomization.
Ventricular premature complex (VPC) evaluated on Holter ElectroCardiogramm (ECG) | three months post-randomization
  VPC burden on Holter ECG performed during the hopsital consultation at three months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BOCHATON, Study Chair — Cardiovascular hospital Louis Pradel; Mathieu KERNEIS, Study Director — Department of Cardiology - Pitié Salpêtrière Hospital
Locations (2):
- France (2):
  - Unité de Soins Intensifs Cardiologiques - Hôpital Cardiovasculaire Louis Pradel, Bron
  - Institut de Cardiologie - APHP Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tschope C, Cooper LT, Torre-Amione G, Van Linthout S. Management of Myocarditis-Related Cardiomyopathy in Adults. Circ Res. 2019 May 24;124(11):1568-1583. doi: 10.1161/CIRCRESAHA.118.313578. PMID 31120823
- [Background] Ammirati E, Cipriani M, Moro C, Raineri C, Pini D, Sormani P, Mantovani R, Varrenti M, Pedrotti P, Conca C, Mafrici A, Grosu A, Briguglia D, Guglielmetto S, Perego GB, Colombo S, Caico SI, Giannattasio C, Maestroni A, Carubelli V, Metra M, Lombardi C, Campodonico J, Agostoni P, Peretto G, Scelsi L, Turco A, Di Tano G, Campana C, Belloni A, Morandi F, Mortara A, Ciro A, Senni M, Gavazzi A, Frigerio M, Oliva F, Camici PG; Registro Lombardo delle Miocarditi. Clinical Presentation and Outcome in a Contemporary Cohort of Patients With Acute Myocarditis: Multicenter Lombardy Registry. Circulation. 2018 Sep 11;138(11):1088-1099. doi: 10.1161/CIRCULATIONAHA.118.035319. PMID 29764898
- [Background] Kyto V, Sipila J, Rautava P. Rate and patient features associated with recurrence of acute myocarditis. Eur J Intern Med. 2014 Dec;25(10):946-50. doi: 10.1016/j.ejim.2014.11.001. Epub 2014 Nov 7. PMID 25468248
- [Background] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965
- [Background] Imazio M, Brucato A, Cemin R, Ferrua S, Maggiolini S, Beqaraj F, Demarie D, Forno D, Ferro S, Maestroni S, Belli R, Trinchero R, Spodick DH, Adler Y; ICAP Investigators. A randomized trial of colchicine for acute pericarditis. N Engl J Med. 2013 Oct 17;369(16):1522-8. doi: 10.1056/NEJMoa1208536. Epub 2013 Aug 31. PMID 23992557